CLINICAL TRIAL: NCT06831331
Title: NUTRA- Nutrition in Rheumatoid Arthritis
Brief Title: Nutrition in Rheumatoid Arthritis
Acronym: NUTRA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NUTRA
Record Dates: First submitted 2025-01-27; First posted 2025-02-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: nutrition; diet; nordic nutrition recommendations; inflammation; metabolomics; cardiovascular risk factors
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant will informed that we test two different diets Care provider will not be informed about which diet the participant consume Outcome will be assessed blinded to which intervention is which
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition recommendations (REC) (Active Comparator): Diet following the Nordic Nutrition Recommendations 2023
  Interventions: Other: REK-diet
- Nutrient rich diet, (RICH) (Active Comparator): Diet rich in nutrients and with high quality protein
  Interventions: Other: RICH-diet

INTERVENTIONS:
Other: REK-diet — Personalized diet- the participants will get individual advice how to adapt their habitual diet to the Nordic Nutrition Recommendations 2023
  Arms: Nutrition recommendations (REC)
Other: RICH-diet — Diet rich in nutrients and with high quality protein
  Arms: Nutrient rich diet, (RICH)

SUMMARY:
Background: Individuals with Rheumatoid Arthritis (RA) often experience persistent symptoms such as pain and stiffness despite modern pharmacological treatments. They also have an increased risk of cardiovascular disease. Elevated risk factors for cardiovascular disease limit the options for symptom-relieving medications, making a reduction in these risk factors highly desirable. Diet has been shown to reduce several of these factors, but the scientific evidence for rheumatoid arthritis is limited, and thus tailored dietary advice is lacking.

Objective: The purpose of the NUTRA study is to evaluate the effect of a diet that follows the updated Nordic Nutrition Recommendations (2023) on disease activity and cardiovascular risk factors in individuals with newly diagnosed RA. Specifically, the study will analyze the impact of the diet on clinically relevant markers such as blood pressure, lipid profile, inflammatory markers, and body composition.

Study Plan: The study will include about 150 patients, and participants will follow a standardized care protocol where, at their three-month visit, they are randomized into either a diet following the Nordic Nutrition recommendations or a Nutrient rich diet. The intervention diets, will be added as a complementary treatment to the medications the patients are already taking. Participants will receive menus, recipes and some foods for three months, followed by self-maintenance of the diet. Clinical markers will be evaluated before the intervention as well as at three and nine months. Artificial intelligence will be used to predict which factors are crucial for achieving the best possible outcomes from dietary treatment.

Significance: The NUTRA study is highly significant as it aims to generate evidence to guide the design of dietary interventions for patients with rheumatoid arthritis. By understanding the potential role of diet in reducing both disease activity and cardiovascular risk, the study may contribute to improved treatment strategies for this challenging patient group.

DETAILED DESCRIPTION:
Study Design and Methodology for NUTRA The NUTRA-trial is a 3-month randomized, controlled, parallel dietary intervention trial. It will compare a personalized healthy diet intervention following the updated Nordic Nutrition Recommendations 2023 to a nutrient rich diet. The Nordic Nutrition Recommendations is evidence based recommendations with focus to limit the dietary risks associated to the burden of disease (specifically ischemic heart disease, type 2 diabetes, stroke and colon and rectum cancers) in the Nordic countries.

Study participants and recruitment: Patients diagnosed with RA in the Gothenburg region and additional sites in Sweden will be recruited for three years. All patients that are diagnosed with RA are "labelled" with "care process RA" in the Healthcare Information Systems (HIS) (for example ELVIS in Region Vastra Gotaland) of Sweden. The investigators will select and invite all patients coded with RA diagnosis by letter within three months from diagnosis. The investigators expect to recruit about 110-150 men and women, likely resulting in about 100-120 participants completing the dietary intervention period and 100 participants the 1 year (i.e. six months after dietary intervention) follow up. Additional sites will be added to increase the recruitment pace if needed. The recruitment pace, compliance, study setup and budget will be evaluated after recruitment and completion of the first 3 months of the study for the first ten participants (during 2025).

Standard care pharmacological treatment: According to the course of medical care most patients diagnosed with RA will start on the first-line treatment (Methotrexate and/or cortisone) immediately after diagnosis. At the three-month clinic visit treatment is evaluated and most patients continue Methotrexate, and some will be offered additional biological treatment. Participants continuing Methotrexate and/or additional biological treatment will be invited to continue in NUTRA-trial.

Data and sample collection: Patients with RA follow a course of medical care. Study baseline (visit 1) will be jointly with the three-month clinical visit, visit 2 with the six-month clinical visit and visit 3 with the 12-month clinical visit. Data will be collected from the clinical visits. In addition, visits before (visit 1) and after (visit 2) the intervention period will include blood and urine collection, clinical phenotype, blood pressure, a 4-day weighed dietary dairy, joint examination, questionnaires (SF-36, HAQ) and physical activity (activity/fitness tracker during the whole period). Visit 1 will also include study information, informed consent, randomization, and a food frequency questionnaire. Patients will be followed up six months after intervention (visit 3) to evaluate if dietary changes persist and for CVD risk factors including lipid patterns.

Assignment: Participants will be randomized (1:1) to either Nordic Nutrition recommendation or Nutrient rich diet intervention at the baseline visit (3 months post diagnosis, visit 1). Randomization will be stratified for site, sex, BMI, and diagnosis (seropositive or negative including both rheumatoid factor (RF) and anticitrullinated protein antibody (ACPA)). To reduce risk of bias, cut-offs for age, diagnosis and block size will be unknown to study personnel that select patients coded with "care process RA" from the system. In addition, block size will be of different sizes, so that risk for allocation bias will be maximally reduced.

Nutrition recommendation: Participants will receive a startup grocery bag and be encouraged to follow the Nordic Recommendations 2023. In addition, a dietitian will provide personalized dietary advice based on the 4-day dietary diary, to improve compliance and to ensure that the participants reach dietary goals.

Nutrient rich diet: Participants will receive a startup grocery bag and be encouraged to consume nutrient rich foods with high protein quality such as meat, dairy and egg, but without menus to support this intake. They will be offered personalized dietary advice after the 12-month clinical visit.

Both groups will wear activity/fitness devices during the intervention period to measure physical activity and will be encouraged to lose weight if overweight. All will also get some general advice regarding a healthy diet, physical activity, and weight within the ordinary care.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed RA (within 3 months) that have started on Methotrexate and/or cortisone treatment. RA is defined according to the criteria from EULAR/American College of Rheumatology (ACR) 2010.
* BMI 18.5-40 kg/m2
* willing to follow the intervention diet

Exclusion Criteria:

* pregnancy
* lactation
* diagnosis for cancer or other life-threatening diseases
* diabetes type 1 and 2
* inflammatory bowel disease or celiac disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Patterns of serum inflammatory markers | 3 months dietary intervention
  Olink Target 96 Inflammation panel will be analysed and multivariate method (OPLS-DA) will be used to evaluate changes in the inflammatory markers between intervention and control.

SECONDARY OUTCOMES:
Remission yes/no | 3 months dietary intervention and at 9 months follow up
  Based on disease activity score -28 joints-erythrocyte sediment rate (DAS28-ESR) and European League Against Rheumatism (EULAR) criteria
Disease activity DAS28-CRP | 3 months dietary intervention and at 9 months follow up
  based on disease activity score -28 joints-c-reactive protein (DAS28-CRP)
Apolipoprotein B100 | 3 months dietary intervention and at 9 months follow up
triacylglycerides | 3 months dietary intervention and at 9 months follow up
high density lipoprotein | 3 months dietary intervention and at 9 months follow up
  HDL
Low density lipoprotein (LDL) | 3 months dietary intervention and at 9 months follow up
total cholesterol | 3 months dietary intervention and at 9 months follow up
Erythrocyte sediment rate (ESR) | 3 months dietary intervention and at 9 months follow up
high sensitive-C-reactive protein (hs-CRP) | 3 months dietary intervention and at 9 months follow up
Corticosteroid use | 3 months dietary intervention and at 9 months follow up
  Participants will note the use of corticosteroids. A decrease could indicate less pain. Changes is also important to adjust for in analysis of effects on inflammation markers.
Physical disability | 3 months dietary intervention and at 9 months follow up
  Based on the questionnaire HAQ THE HEALTH ASSESSMENT QUESTIONNAIRE (HAQ) DISABILITY INDEX (DI) There are 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). Total score is divided to the number of categories and the range of the index is thus 0-3p.
Quality of life (RAND-SF36) | 3 months dietary intervention and at 9 months follow up
  Self-reported quality of life based on the questionnaire 36-Item Short Form Survey Instrument (SF-36) from RAND (Research and Development- non profit organisation). It taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Scale is 0-100. Higher score indicates better quality of life.
Disease activity score DAS28-ESR | 3 months dietary intervention and at 9 months follow up
  Disease activity score based on 28 joints and erythrocyte sediment rate (ESR)

OTHER OUTCOMES:
Body mass index (BMI) | 3 months dietary intervention and at 9 months follow up
  Patients are not advised to actively try to loose weight, but do not have to try to keep their weight either. BMI will be a descriptive measure.
Body composition | 9 months follow up
  Dual x ray absorptiometry (DXA) at baseline and 9 months Descriptive/for adjustment and relative to both diet and eventual changes in physical activity
Patterns of metabolites | 3 months dietary intervention
  Metabolites analysed by NMR or LC-MS/GC-MS for metabolomics studies (changes in patterns of metabolites). This outcome will mainly be used to evaluate compliance to the intervention diet. Metabolite patterns will be compared by multivariate methods such as OPLS-DA. This outcome will also be used at baseline for descriptives of the participants i.e. habitual lifestyle and diet.
European League Against Rheumatism (EULAR) criteria for disease activity | 3 months dietary intervention and at 9 months follow up
  Based on Disease Activity Score -28 joints -Erythrocyte sediment rate. This can be used to classify patients as good, moderate or non-responders, using the individual amount of change in the DAS and the DAS value (low, moderate, or high) reached. Classes can be used to explore differences in baseline metabolomics, gut microbiota and body composition.
Differences in changes in fatty acid patterns in plasma | 3 months dietary intervention
  Fatty acids will be analysed in plasma and patterns of fatty acids will be analysed and changes in fatty acid patterns during intervention and control will be compared with multivariate methods as a marker for compliance to the diets.
Differences in changes in fatty acid patterns in erythrocytes | 3 months dietary intervention
  Fatty acids will be analysed in erythrocytes and changes in fatty acid patterns during intervention and control will be compared with multivariate methods as a marker for compliance to the diets.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinisk Reumatologiskt Forskningscentrum, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Not eligible according to Swedish law

REFERENCES:
- See also: Information about the study for presumptive participants- IN SWEDISH — https://www.gu.se/medicin/delta-i-studie-om-kost-vid-ledgangsreumatism
- See also: About this study and previous studies within the same research area- IN SWEDISH — https://www.gu.se/forskning/kost-vid-kroniska-inflammatoriska-sjukdomar